CLINICAL TRIAL: NCT05854446
Title: Navigating the Challenges of Myofascial Pain Syndrome in Turkey: A Delphi Methodology Study on Patient Journey, Disease Burden, and Unmet Diagnosis and Treatment Needs
Brief Title: Delphi Study on Myofascial Pain Syndrome Challenges in Turkey: Patient Journey, Burden, Diagnosis & Treatment Needs.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Uskudar State Hospital (Other Government)
Responsible Party: Principal Investigator, Mustafa Hüseyin Temel, Principal Investigator, Uskudar State Hospital
Other Study IDs: MPS1
Record Dates: First submitted 2023-05-02; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Myofascial Pain Syndrome
Keywords: Disease burden; Delphi methodology; Patient journey; Myofascial Pain Syndrome; Quality of life
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthcare Experts: Experts with diverse backgrounds in healthcare and pain management.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — In this survey, The experts will be asked open-ended questions based on the literature research and patient surveys carried out by the researchers in the first round to identify key themes related to myofascial pain syndrome, including the disease burden, patient journey, and unmet diagnosis and treatment needs. In subsequent rounds, the experts will rate the importance of each theme and provide additional feedback.

SUMMARY:
Myofascial pain syndrome is a chronic pain disorder that affects many people in Turkey. This research study aims to explore the challenges faced by patients with myofascial pain syndrome in Turkey, including the disease burden, patient journey, and unmet diagnosis and treatment needs. The study will utilize the Delphi methodology, which involves gathering input from a panel of experts over multiple rounds to achieve consensus on the topic. The results of this study will shed light on the current state of myofascial pain syndrome management in Turkey and provide insights into the areas where improvements can be made.

DETAILED DESCRIPTION:
The study will use a Delphi methodology to investigate the challenges faced by patients with myofascial pain syndrome in Turkey. A panel of 20 experts with diverse backgrounds in healthcare and pain management will be selected. The study will be conducted in three rounds, with the first round consisting of open-ended questions to identify key themes related to the disease burden, patient journey, and unmet needs. In the second round, experts will rate the importance of each theme, and in the third round, they will review the results of the previous round and provide additional feedback. Data will be analyzed using content analysis and descriptive statistics to identify the areas of consensus and divergence among the experts.

ELIGIBILITY:
Inclusion Criteria:

* Being an expert on healthcare.
* Giving consent.

Exclusion Criteria:

* Not giving consent.
* Any disorder or condition that may negatively affect reading, comprehension, and form filling.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A panel of 20 experts from diverse backgrounds in healthcare and pain management.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Identification of areas of agreement and disagreement among experts. | 1 month
  Data will be analyzed using content analysis and descriptive statistics to identify the areas of consensus and divergence among the experts.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa H Temel, M.D., Principal Investigator — Uskudar State Hospital

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will be shared by the corresponding author upon reasonable request.